CLINICAL TRIAL: NCT05223296
Title: LigaSure or Diathermy Excision of III-IV Degree Pile? A Single-institution Experience: Randomized Control Trials
Brief Title: LigaSure or Diathermy Excision of III-IV Degree Pile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jabir Ibn Hayyan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pile
Record Dates: First submitted 2022-01-04; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Pile
Keywords: ligaSure; pile; diathermy; hamemorrdectomy; grade II-IV pile
MeSH Terms: conditions — Hemorrhoids; Fever

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I LigaSure (n=100) (Active Comparator): 100 patients subjected to LigaSure pile excision
  Interventions: Device: Compare between two procedure for II-IV degree pile excision
- Group II Conventional diathermy (n=108) (Active Comparator): 108 patients subjected to conventional diathermy for grade IV pile excision
  Interventions: Device: Compare between two procedure for II-IV degree pile excision

INTERVENTIONS:
Device: Compare between two procedure for II-IV degree pile excision — LigaSure or diathermy excision of III-IV degree pile?

SUMMARY:
Abstract:

Introduction:

Pile excision is frequently associated with post-operative pain and prolong hospital stay. A modern technique performed with LigaSure appears to be mainly effective in large pile tissue removal is required. The study compares LigaSure pile excision with diathermy for the treatment of III-IV degree pile.

Patients and Methods:

208 patients with pile III or IV degree randomized into 2 groups. Group one LigaSure and group two diathermy. The study evaluates the mean post-operative time, post-operative pain, discharge date, time return to usual works early and late complication. All patient followed-up for range (12-24) months.

Results:

108patient treated by diathermy, 100 by LigaSure. The mean operative time significantly shorter in LigaSure, post-operative pain disappears earlier in LigaSure than diathermy. The time return to work less in LigaSure, while no difference in hospital stay and post-operative complications.

Conclusions:

LigaSure is effective procedure when large degree III or VI pile excised. The procedure enhances to use LigaSure as treatments of choice for class III-IV pile, even it is more expensive than diathermy operation.

DETAILED DESCRIPTION:
Surgery remains the mainstay in patients with symptomatic pile grades III and IV. The usual operation by Milligan-Morgan and Ferguson is still most used and effective for symptomatic grades IV and some of grade III. The two procedures get mimicked, like blood loss and postoperative pain, which cause prolonged hospital stay. Rapid wound healing permits the early return to usual works and day activity . Many articles seek the best treatments of piles published in recent years and modern device the procedures trials to overcome the haemorrhoidectomy complication.: like stapling, laser, doppler-guided vessels ligation with different principles aimed at excisional surgery. The LigaSure system vessels sealed were introduced newly in [6] as a tool for treatments of piles. It is a bipolar electro-thermal device; it offers both radiofrequency and pressure. Blood vessels seal up to 7mm in diameter and create energy according to the tissue impendence and confined 2 mm thermal injury over operation site. The limited thermal injury spread decreases the anal spasm and permits bloodless surgery to decrease postoperative pain and promote rapid healing. So the operation is recommended as an ideal procedure because of the significant less tissue trauma . The objective of some randomized trials to estimate the advantage of the LigaSure approach over the conventional diathermy approaches. in spite of the favourite toward the LigaSure, the conclusion gets some uncertainly regarding the cost of using disposable device although an overall favourable trend exists toward LigaSure, conclusions are not univocal and definitive; this creates some uncertainty, also considering the increasing cost for the use of the disposable device so essential to compare our study with another centres to emphasis the true advantage present. The debate is the "gold standard" for III degrees. There are large agreements that Milligan-Morgan and Ferguson are the most effective in IV degree pile . Ortiz mentions that stapled procedure is ineffective for curing itching in an IV degree pile . So the diathermy pile excision continues as an effective therapy for the symptomatic, irreducible and prolapsed pile. The designed study to estimate the LigaSure procedures as effective as conventional diathermy in all grades IV and III with less pain, less blood loss and when we need large tissue excision needed.

ELIGIBILITY:
Inclusion Criteria:

III-IV degree pile Prolapsed, irreducible pile

Exclusion Criteria:

I-II degree pile Internal pile

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2020-01-19 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
postoperative pain,complication, time return to home activity | two years
  LigaSure better than diathermy in grade II-IV pile excision

CONTACTS AND LOCATIONS:
Overall Officials: Adel Al-Mayely, Ph.D., Study Director — Jabir Ibn Hayyan Medical University
Locations (1):
- Samer Al-Hakkak, Najaf, An Najaf, Iraq

IPD SHARING:
Plan to Share IPD: No